CLINICAL TRIAL: NCT04050423
Title: Investigation of Ultrasound Imaging and Spectroscopy for Characterizing Breast Masses
Status: Recruiting | Type: Observational
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Dr. Gregory Czarnota, Radiation Oncologist and Clinician Scientist, Sunnybrook Health Sciences Centre
Other Study IDs: 232-2014
Record Dates: First submitted 2019-07-22; First posted 2019-08-08 (Actual); Last update posted 2023-12-14 (Actual); Status verified 2023-12

CONDITIONS: Breast Cancer
Keywords: Ultrasound; Spectroscopy; Characterization
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Our objective in this study is to identify an optimal set of quantitative ultrasound parameters that can be used, non-invasively, to characterize breast masses with high accuracy, as determined histopathologically. Breast cancer is the most frequent form of non-epithelial cancer diagnosed in women, with approximately 1.5 million new cases diagnosed annually worldwide. Accurate diagnosis and characterization of disease play an important role in therapy planning for breast cancer treatment. Currently, the gold standard method of tumour diagnosis is pathological examination of core biopsy specimens. However, the invasive core biopsies can cause post-surgical complications. Besides, some lesions require repeat biopsy due to sampling errors during the initial biopsy. Also X-ray mammography and ultrasound B-mode images, which are used by radiologists for breast examination, lack reliable information about micro-structural properties of tissues. There is an urgent need of a non-invasive imaging modality that can provide rapid and quantitative information for breast tumour characterization, in real time and at the patient bed. The main goal, as described above, is to select the best quantitative ultrasound parameters that can facilitate breast cancer characterization, non-invasively.

DETAILED DESCRIPTION:
This project is an observational/early validation study in human subjects that will use ultrasound imaging and spectroscopy to characterize suspected breast cancers. Patients will be imaged with ultrasound, and the acquired data will be analyzed using quantitative ultrasound techniques, in conjunction with textural analysis on generated parametric images. Results of quantitative ultrasound data analysis for these breast lumps will be compared to and correlated with their histopathological characteristics from pathology reports on core biopsy specimens, surgery reports, or radiology reports, available from patient charts. From this data we will potentially estimate the best hybrid ultrasound-based biomarker that can characterize suspected breast cancers, noninvasively.

ELIGIBILITY:
Inclusion Criteria:

1. Women or men with suspected breast cancer
2. Patients should have the ability to understand and the willingness to sign a written Informed consent document.

Exclusion Criteria:

1. Patients who have had chemotherapy, radiotherapy, or major surgery within 4 weeks prior to registering in the study or those who have not recovered from adverse events due to agents administered more than 4 weeks prior to registration
2. Receiving any other investigational agents
3. Any condition that is unstable or could jeopardize the safety of the patient and their compliance in the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Both men and women and members of all races and ethnic groups are eligible for this trial.
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2014-09-23 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2029-09 (Estimated)

PRIMARY OUTCOMES:
Select the best quantitative ultrasound parameters that can facilitate breast cancer characterization, non-invasively | Up to 5 years
  Correlate quantitative ultrasound parameters obtained using spectroscopic techniques, in conjunction with textural analysis on generated parametric images, to the histopathological characteristics from pathology reports on core biopsy specimens, surgery reports, or radiology reports.

SECONDARY OUTCOMES:
Results of ultrasound-based breast cancer characterization and clinical outcomes. | Up to 5 years
  Correlating the results of ultrasound-based breast cancer characterization.

CONTACTS AND LOCATIONS:
Overall Officials: Gregory J Czarnota, PhD, MD, Principal Investigator — Sunnybrook Health Science Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada